CLINICAL TRIAL: NCT06782854
Title: Understanding the Role of Large Extracellular Vesicles in Lymphomas and Lymphoproliferative Disorders: the "Off the Beaten Track" Liquid Biopsy - A Prospective Monocentric in Vitro Study on Human Tissues
Brief Title: Understanding the Role of Large Extracellular Vesicles in Lymphomas and Lymphoproliferative Disorders: the "Off the Beaten Track" Liquid Biopsy
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: EVs-Lympho; RC-2024-2790168 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2024-12-30; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Diffuse Large B-Cell Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma(MZL); Mycosis Fungoides; Chronic Lymphocytic Leukemia; Hairy Cell Leukemia (HCL); T Cell Lymphoma; Multiple Mieloma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Mycosis Fungoides; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Lymphoma, T-Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the role of extracellular vesicles as diagnosic and prognostic biomarkers in patients with lymphomas or lymphoproliferative disorders. In particular, circulating extracellular vesicles, thanks to their cargo of proteins, lipids, and nucleic acids, play a role in the communication between cells. Since it has been described that these vesicles are able to influence also immune cells, the study of their functions may lead to the discovery of new mechanisms underlying this type of diseases.

DETAILED DESCRIPTION:
It is a 3-year monocentric in vitro study on human tissue. 50 patients with aggressive and indolent Non-Hodgkin Lymphomas (Diffuse Large B-Cell Lymphoma (DLBCL; Group A; n=10), Follicular Lymphoma (FL; Group B; n=10), Marginal Zone Lymphoma (MZL; Group C; n=10), Peripheral T-Cell Lymphoma (PTCL; Group D; n=10), Mycosis Fungoides (MF; Group E; n=10)), and patients with Chronic Lymphocytic Leukaemia (CLL; N=10; Group F; n=10), Hairy Cell Leukemia (HCL; Group G; n=10), and Multiple Myeloma (MM; N=10; Group H; n=10) will be enrolled over a period of 24 months. Follow-up: 12 months. Patients will be enrolled at the Complex Operative Unit of Haematology-IRCCS Azienda Ospedaliero-Universitaria di Bologna. The peripheral blood samples of patients (40 ml) will be collected only at diagnosis within normal clinical practice, outside of clinical study protocols, and following the treatment guidelines in use at the Centre. The analysis of the samples will be performed at the Unità Operativa Complessa di Ematologia-IRCCS Azienda Ospedaliero-Universitaria di Bologna in collaboration with the Istituto Romagnolo per lo Studio dei Tumori 'Dino Amadori' - IRST IRCCS and with the University of Perugia.

ELIGIBILITY:
Inclusion criteria for patients:

* Age ≥ 18 years.
* Patients with WHO 2017-defined diagnosis of indolent and aggressive Non-Hodgkin Lymphoma (specifically Diffuse Large B-Cell Lymphoma, Follicular Lymphoma, Marginal Zone Lymphoma, Peripheral T-Cell Lymphoma, Mycosis Fungoides) or Chronic Lymphocytic Leukemia or Hairy Cell Leukemia or Multiple Myeloma.
* Signed informed consent.

Exclusion criteria for patients:

- Concomitant secondary neoplasia.

Inclusion criteria for healthy donors:

* Age ≥ 18 years.
* Signed informed consent.

Exclusion criteria for healthy donors:

- Healthy donors with neoplasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at diagnosis (Diffuse Large B-Cell Lymphoma, Follicular Lymphoma, Marginal Zone Lymphoma, Peripheral T-Cell Lymphoma, Mycosis Fungoides, Chronic Lymphocytic Leukemia, Hairy Cell Leukemia, Multiple Myeloma) will be enrolled over a 24 month period. Follow-up 1 year.
  Sex/age matched healthy donors will be recruited for peripheral blood collection among volunteers of a no profit organization called Bologna AIL.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2024-11-17 (Actual)

PRIMARY OUTCOMES:
Extracellular vesicle characterization | 2 years
  Comparison of concentration (particles/ml), phenotype, and cargo of extracellular vesicles from patients and healthy donors.
Validation of extracellular vesicles as biomarker | 2 years
  Correlation of extracellular vesicles' characterization results with biomarkers of disease aggressiveness and short-term response to standard therapy.

SECONDARY OUTCOMES:
Functional effects of extracellular vesicles | 2 years
  Comparison of functional effects of extracellular vesicles from patients and healthy donors on selected immune cells. The isolated vesicles will be used to treat the immune cells (T cells, B cells, monocytes) to evaluate viability, phenotype, migration ability, and inflammatory cytokine production of the target cells.

OTHER OUTCOMES:
Extracellular vesicles' cell of origin | 1 years
  Correlation of extracellular vesicles' phenotype with the corresponding cells of origin.

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Catani, PhD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy